CLINICAL TRIAL: NCT04380012
Title: Pyrotinib Maleate With or Without Trastuzumab in the Treatment of HER2-positive Advanced Colorectal Cancer: a Multicenter Clinical Trial
Brief Title: A Clinical Study of Pyrotinib in Patients With HER2-positive Advanced Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Zhejiang Cancer Hospital (Other); Zhejiang Provincial People's Hospital (Other); First Affiliated Hospital of Zhejiang University (Other); Sir Run Run Shaw Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IR2019001210
Record Dates: First submitted 2020-02-04; First posted 2020-05-08 (Actual); Last update posted 2021-07-15 (Actual); Status verified 2021-02

CONDITIONS: Colorectal Cancer
Keywords: HER2; Advanced Colorectal Cancer; Pyrotinib
MeSH Terms: conditions — Colorectal Neoplasms | interventions — pyrotinib; Trastuzumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single drug group (Experimental): Pyrotinib: 400 mg, po, qd, 21d for a treatment cycle
  Interventions: Drug: Pyrotinib
- Dual-targeted drug group (Experimental): Pyrotinib: 400 mg, po, qd, 21d for one treatment cycle; Trastuzumab: first dose 8 mg/kg, then 6 mg/kg, iv, q3w, 21d for one treatment cycle
  Interventions: Drug: Pyrotinib in combination with trastuzumab

INTERVENTIONS:
Drug: Pyrotinib — Pyrotinib as interventions were used in patients with HER2-positive advanced colorectal cancer
  Arms: Single drug group
Drug: Pyrotinib in combination with trastuzumab — Pyrotinib in combination with trastuzumab as interventions were used in patients with HER2-positive advanced colorectal cancer
  Arms: Dual-targeted drug group

SUMMARY:
To Observe the Efficacy and Safety of Pyrotinib Maleate in Patients With HER2-positive Advanced Colorectal Cancer

DETAILED DESCRIPTION:
This study is an investigator-initiated, open-label, two-cohort phase II trial, assessing the objective response rate (ORR) of pyrotinib monotherapy (Cohort 1) or in combination with trastuzumab (Cohort 2), in HER2-positive advanced colorectal cancer.

HER2 positivity is centrally established by immunohistochemistry (IHC) and silver in situ hybridization (SISH). To be HER2 eligible the original tumor, or the biopsied metastasis (whichever is last available), must be IHC 3+ or 2+ in more than 50% of cells, confirmed by SISH or fluorescence in situ hybridization (FISH) with a HER2:CEP17 ratio ≥ 2.0. For IHC a positive staining (3+) is defined as an intense membrane staining which can be circumferential, basolateral, or lateral of the tumor cells.

ELIGIBILITY:
Inclusion Criteria:

* 1. Aged 18-75 years, male or female;
* 2. ECOG performance status 0-2;
* 3. Recurrent/metastatic advanced colorectal cancer diagnosed by histology or cytology;
* 4. Patients who progressed on or were intolerable to standard therapy, or those who refused chemotherapy;
* 5. At least one measurable lesion according to RECIST v1.1;
* 6. HER2 positivity (including amplification, mutation, and overexpression) detected by clinically recognized methods (including PCR, FISH, immunohistochemistry, and NGS), and the data obtained by NGS at the pathology department of hospital or qualified gene testing organization could be accepted;
* 7.The functional level of the major organs must meet the following requirements (no blood transfusion within 2 weeks prior to screening, no use of leukocytes- or platelet-raising drugs):

  1. Blood routine: neutrophils (ANC) ≥ 1.5 × 10^9 / L; platelet count (PLT) ≥ 90 × 10^9 / L; hemoglobin (Hb) ≥ 90 g / L;
  2. Blood biochemistry: total bilirubin (TBIL) ≤ upper limit of normal (ULN); alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2 × ULN（Patients with liver metastases were ≤5 × ULN）;
  3. Cardiac color doppler ultrasound: left ventricular ejection fraction (LVEF) ≥ 55%;
  4. 12-lead electrocardiogram: The QT interval corrected by the Fridericia method (QTcF) < 470 msec;
* 8. Sign the informed consent and agree to collect the clinical efficacy and information of the patient.

Exclusion Criteria:

* 1. The presence of third interstitial effusion (such as a large amount of pleural fluid and ascites) that cannot be controlled by drainage or other methods makes it impossible to evaluate the clinical treatment effect;
* 2. History of substance abuse and cannot be cured or with mental disorders;
* 3. Pregnant or lactating women; patients with fertility who are unwilling or unable to use effective contraception;
* 4. Severe concomitant disease, or unsuitable to participate in this study decided by the investigator.
* 5. Prior use of pyrotinib.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-12-17 (Actual); Primary Completion 2021-12-17 (Estimated); Study Completion 2022-06-17 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | Approximately 24 months
  The proportion of patients with complete response or partial response according to RECIST v1.1.

SECONDARY OUTCOMES:
Disease Control Rate | Approximately 24 months
  The proportion of patients with complete response, partial response or stable disease according to RECIST v1.1.
Progression-Free Survival | Up to 2 years
  Time from the initiation of treatment to disease progression or any-cause death.
Overall Survival | Up to 2 years
  Time from the initiation of treatment to any-cause death.
Duration of Response | Approximately 24 months
  Time from complete response or partial response to disease progression or any-cause death.
The Incidence of Adverse Events | From the first drug administration to within 28 days for the last treatment
  Adverse Events and Serious Adverse Events were graded according to the NCI-CTCAE V5.0.

CONTACTS AND LOCATIONS:
Locations (1):
- The Second Affiliated hospital of Zhejiang University School of Medical, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided
The data were Shared with the sub-center, and the preliminary efficacy results were to be submitted to the tumor conference